CLINICAL TRIAL: NCT00979277
Title: Transcriptomal and Molecular Characterization of Tumor Associated Monocytes / Macrophages in Human Cancers
Brief Title: Transcriptomal and Molecular Characterization of Tumor Associated Monocytes/Macrophages in Human Cancers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Haematology-Oncology, Alvin Wong, Senior Consultant, National University Hospital, Singapore
Other Study IDs: MC03/17/07
Record Dates: First submitted 2009-09-15; First posted 2009-09-17 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Tumor; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Recent studies from both human and mice cancer models have demonstrated a crucial role for monocytes/macrophages in contributing to cancer progression and disease prognosis. However, since each cancer subtypes is associated with a unique tumor microenvironment in terms of its anatomical location, cytokine/chemokine profiles and stromal components, the functional contribution of tumor infiltrating cells such as the monocytes/macrophages can be equally diverse, depending on the type of cancer. Therefore to obtain a global understanding of the role of host immune cells in cancer progression, it is necessary to accurately characterize these cells in the context of the tumor microenvironment for several cancer subtypes rather than a single cancer. In view of this, this pilot proposal aims to carryout a systems approach in characterizing the functional phenotype of monocyte/macrophage lineage in 4 diverse human cancer types [e.g., Colorectal Cancer, Nasopharyngeal carcinoma, Hepatocellular (liver) cancer and Renal cell carcinoma (kidney cancer)] and the molecular basis of tumor-induced immunosuppression in each of these conditions. Besides providing a global view of the host innate immunity and its molecular basis in these human cancer, the outcome of this investigation will be crucial in defining the scopes of specific immunotherapy strategies to overcome tumor-induced immunosuppression and induce monocyte/macrophage-mediated antitumor response.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the inclusion criteria to participate in this study:

* Diagnosed NPC, RCC, HCC or colorectal cancer patients. (Preoperative histologic diagnosis is not required for RCC and HCC.)
* All stages of disease are eligible.
* Adult patients above 21.
* Ability to provide informed consent.

Exclusion Criteria:

Subjects meeting any of the exclusion criteria at baseline will be excluded:

* Active infection.
* Immunocompromised or other active immune disorders.
* Have received chemotherapy or other immunomodulating therapy in the past 6 months.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 15 subjects from each tumor type. (NUH: NPC 15, CRC 15, RCC 7, HCC 8. AH: HCC 7,TTSH: RCC 8)
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Balkwill F, Charles KA, Mantovani A. Smoldering and polarized inflammation in the initiation and promotion of malignant disease. Cancer Cell. 2005 Mar;7(3):211-7. doi: 10.1016/j.ccr.2005.02.013. No abstract available. PMID 15766659
- [Background] Balkwill F, Mantovani A. Inflammation and cancer: back to Virchow? Lancet. 2001 Feb 17;357(9255):539-45. doi: 10.1016/S0140-6736(00)04046-0. PMID 11229684